CLINICAL TRIAL: NCT02637011
Title: Influence of Quality of Care and Individual Patient Characteristics on Quality of Life/ Return to Work in Survivors of the Acute Respiratory Distress Syndrome (ARDS): Prospective, Observational, Multi-centre Cohort Study
Brief Title: Surviving ARDS: The Influence of Quality of Care and Individual Patient Characteristics on Quality of Life
Acronym: DACAPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Regensburg (Other)
Collaborators: University of Regensburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Bein M.A., Principal Investigator, University Hospital Regensburg
Other Study IDs: 01GY1340
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: acute respiratory distress syndrome; intensive care medicine; critical illness; long-term outcomes; quality of life; return to work; quality of care
MeSH Terms: conditions — Respiratory Distress Syndrome; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the DACAPO study ("Surviving ARDS: the influence of quality of care and individual patient characteristics on quality of life") is to investigate the role of quality of care and individual patient characteristics on quality of life and return to work in survivors of ARDS (acute respiratory distress syndrome). It is hypothesized that higher quality of care is associated with better health-related quality of life and a higher rate of return to work among survivors.

A prospective, observational, multi-centre patient cohort study is performed in Germany, using hospitals from the "ARDS Network Germany" as the main recruiting centres. It is envisaged to recruit 2400 patients into the DACAPO study and to analyze a study population of 1500 survivors. They will be followed up until 12 months after discharge from hospital. Quality of care will be assessed as process quality, structural quality and volume at the institutional level. The main outcomes (health related quality of life and return to work) will be gathered by self-report questionnaires. Further data assessment includes general medical and ARDS-related characteristics of patients as well as sociodemographic and psycho-social parameters. Multilevel hierarchical modelling will be performed to analyse the effects of quality of care and individual patient characteristics on outcomes, taking the cluster structure of the data into account.

DETAILED DESCRIPTION:
Design Patients will be included in the study at the beginning of ICU stay in a participating hospital (t0) and survivors will be followed over a period of 12 months after discharge from ICU. If patients have been treated before in a referring hospital, a retrospective assessment of their health status during their stay in this hospital and during inter-hospital transport will be performed. Four follow-up measurements (at discharge from ICU as well as 3, 6 and 12 months after discharge) will be performed on individual patient level.

Sample & Recruitment Hospitals of the "ARDS Network Germany" and other hospitals which provide care for patients with ARDS were invited to participate in the study.

It is envisaged to screen 2600 patients for the presence of ARDS and to include 2400 patients as members of the source population. An in-hospital mortality rate of 30% is assumed; therefore, we expect to analyze a study population of 1500 patients at t1 (discharge from ICU). For each follow-up-assessment (t2-t4: 3 months, 6 months, 12 months after discharge), loss-to-follow-up rates due to death, withdrawal of consent or other reasons are estimated to be about 10%, resulting in slightly more than 1000 patients at 12-months-follow-up.

Measurements The main predictor is quality of care provided in the ICUs of the participating hospitals. The following main indicators were chosen: qualification of physicians, implementation of routine daily multiprofessional ward rounds with documentation of daily therapy goals, number of ventilated patients per, and membership of the hospital in the "ARDS Network Germany". All quality indicators will be assessed by questionnaire at the institutional level.

Main outcome measures of the DACAPO study are HRQoL and return to work among survivors of ARDS (see study outcomes).

Moderating variables are gender, socio-economic status, prevalent and incident psychopathological symptoms (PHQ-D, PTSS-14) and the availability of social support (F-SozU K-14).

Additional variables comprise general medical ICU parameters (e.g. comorbidity, prognostic scores (SAPS (Simplified Acute Physiology Score) II, SAPS III ) and an organ dysfunction score (SOFA (Sequential Organ Failure Assessment score)) and parameters relating to ARDS (e.g. cause and severity) and its treatment (e.g. ventilation parameters, use of supportive care measures, critical events (hypoglycaemia, hypoxia)) as well as socio-demographic and psycho-social characteristics.

Additionally, costs will be assessed as direct costs in terms of treatment costs at the ICU.

Data Sources and Data Collection Patients's general medical characteristics and medical data relating to ARDS and its treatment will be assessed during ICU stay and gathered through electronic case report forms (eCRFs). Data on the direct costs of treating patients with ARDS in the ICU will be gathered from hospital records. A 12-months mortality follow-up will be performed. Local municipal population registries will be contacted to obtain data on mortality at the patient level.

At baseline, caregivers will provide proxy report of patients' socio-demographic data, at follow-ups (discharge from ICU, 3 months, 6 months, 12 months), patients themselves will complete self-report questionnaires on socio-demographic and psycho-social characteristics as well as on the main outcome measures.

Data on indicators of quality of care will be assessed through questionnaires administered to the directors of the hospitals/ICUs.

Data Management The open source software OpenClinica, version 3.1, will be used for electronic data collection and data management. eCRFs will be used for data entry. A continuous assessment of data quality will be performed by exporting data sets to statistical packages to run further error and plausibility checks. Data from paper-pencil-questionnaires completed by patients will be entered into the database twice in order to ensure high data quality.

Statistical Analysis A linear multilevel regression model will be fitted both for the physical and the mental component summary score of the SF-12. A non-parametric multilevel regression model will be used for the outcome "return to work". The modelling procedure will be applied to each of the operationalizations of the predictor "quality of care".

All analyses will be carried out using SAS 9.4 software and STATA version 12 software.

ELIGIBILITY:
Inclusion Criteria:

* ARDS according to the criteria of the Berlin-Definition:

  i) Acute onset within one week, ii) bilateral pulmonary infiltrates (chest imaging), iii) respiratory failure not fully explained by cardiac failure or fluid overload.
* informed consent provided by the patient or the legal guardian
* 18 years old or older

Exclusion Criteria:

* no ARDS
* no informed consent provided by the patient or the legal guardian
* younger than 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected of patients with ARDS treated at intensive care units of the participating hospitals. Participating hospitals are members of the ARDS Network Germany or other hospitals which agreed to take part in the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life, measured by the Short-Form 12-item Health-Survey (SF-12) | 3 months, 6 months, 12 months after discharge from the ICU
  change from baseline (discharge from the ICU) to 3 months, 6 months and 12 months, respectively.

SECONDARY OUTCOMES:
return to work | 3 months, 6 months, 12 months after discharge from the ICU
  Assessment by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bein, Prof. Dr., Principal Investigator — University Hospital Regensburg, Germany
Locations (3):
- Germany (3):
  - Universitätsmedizin Charite, Berlin, State of Berlin
  - Universitätsmedizin Göttingen, Göttingen
  - Klinik für Intensivmedizin, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blecha S, Zeman F, Rohr M, Dodoo-Schittko F, Brandstetter S, Karagiannidis C, Apfelbacher C, Bein T; DACAPO study group. Association of analgosedation with psychiatric symptoms and health-related quality of life in ARDS survivors: Post hoc analyses of the DACAPO study. PLoS One. 2022 Oct 21;17(10):e0275743. doi: 10.1371/journal.pone.0275743. eCollection 2022. PMID 36269731
- [Derived] Apfelbacher C, Brandstetter S, Blecha S, Dodoo-Schittko F, Brandl M, Karagiannidis C, Quintel M, Kluge S, Putensen C, Bercker S, Ellger B, Kirschning T, Arndt C, Meybohm P, Weber-Carstens S; DACAPO study group; Bein T. Influence of quality of intensive care on quality of life/return to work in survivors of the acute respiratory distress syndrome: prospective observational patient cohort study (DACAPO). BMC Public Health. 2020 Jun 5;20(1):861. doi: 10.1186/s12889-020-08943-8. PMID 32503583
- [Derived] Blecha S, Brandl M, Zeman F, Dodoo-Schittko F, Brandstetter S, Karagiannidis C, Bein T, Apfelbacher C; DACAPO Study Group. Tracheostomy in patients with acute respiratory distress syndrome is not related to quality of life, symptoms of psychiatric disorders or return-to-work: the prospective DACAPO cohort study. Ann Intensive Care. 2020 May 6;10(1):52. doi: 10.1186/s13613-020-00671-x. PMID 32377963
- [Derived] Blecha S, Brandstetter S, Dodoo-Schittko F, Brandl M, Graf BM, Bein T, Apfelbacher C. Acceptability of a German multicentre healthcare research study: a survey of research personnels' attitudes, experiences and work load. BMJ Open. 2018 Sep 24;8(9):e023166. doi: 10.1136/bmjopen-2018-023166. PMID 30249633
- [Derived] Dodoo-Schittko F, Brandstetter S, Brandl M, Blecha S, Quintel M, Weber-Carstens S, Kluge S, Kirschning T, Muders T, Bercker S, Ellger B, Arndt C, Meybohm P, Adamzik M, Goldmann A, Karagiannidis C, Bein T, Apfelbacher C; DACAPO Study Group. German-wide prospective DACAPO cohort of survivors of the acute respiratory distress syndrome (ARDS): a cohort profile. BMJ Open. 2018 Apr 4;8(4):e019342. doi: 10.1136/bmjopen-2017-019342. PMID 29622574
- [Derived] Blecha S, Dodoo-Schittko F, Brandstetter S, Brandl M, Dittmar M, Graf BM, Karagiannidis C, Apfelbacher C, Bein T; DACAPO Study Group. Quality of inter-hospital transportation in 431 transport survivor patients suffering from acute respiratory distress syndrome referred to specialist centers. Ann Intensive Care. 2018 Jan 15;8(1):5. doi: 10.1186/s13613-018-0357-y. PMID 29335831